CLINICAL TRIAL: NCT02677909
Title: Computer-Aided, Non-Invasive, Acoustic Gastrointestinal Surveillance (AGIS) in ICU Patients
Status: Withdrawn | Type: Observational
Why Stopped: Did not receive sensors from device company and did not initiate enrollment.
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Matthew Bloom, Assistant Professor of Surgery, Cedars-Sinai Medical Center
Other Study IDs: 01-2016
Record Dates: First submitted 2016-02-05; First posted 2016-02-09 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Critical Illness
Keywords: Parenteral Nutrition; Critical Care
MeSH Terms: conditions — Critical Illness; Hyperphagia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: AEGIS (Automated Evaluation of Gastrointestinal Symptoms) — Will place device on admission to SICU. Measure bowel sounds and await bowel function

SUMMARY:
In this study, the investigators aim to conduct a pilot test of the AbStats device. The v2.0 prototype is a low-profile set of sensors that fits externally around the abdomen and is embedded with specialized wireless sensors. The device continuously, safely, and comfortably monitors intraabdominal acoustic signals, and stores the data in a HIPAA compliant software system.

The investigators will focus this trial on a high-impact inpatient population: ileus in the surgical critical care unit. The investigators will compare the device's signal profiles in patients with ileus vs those who tolerate feeding without high gastric feed residual. Our study will have the following specific aims:

Specific Aim #1: To measure the sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) of initiation day ("PID 0") AGIS signals in predicting PID #1 feeding failure. Specific Aim #2: Among patients tolerating feeds on PID #1, to measure the sensitivity, specificity, PPV, and NPV of AGIS in predicting feeding failure on subsequent icu days.

DETAILED DESCRIPTION:
The AGIS device consists of two acoustic sensors placed on the abdomen to "hear" all segments of the abdominal cavity. Other sensor configurations are possible as needed. Initial testing of this device was conducted at UCLA and VA-Wadsworth under separate IRB approval; however, at this time, all remaining human subjects will be enrolled at CSMC only. We will collect AGIS data in patients undergoing GI abdominal surgery on the day of surgery and throughout their inpatient hospital course.

We will recruit patients who are already scheduled to undergo GI abdominal surgery. The AbStats/AGIS system will be utilized to measure and analyze bowel sounds and correlate with clinical findings. We will exclude subjects who cannot consent, have cognitive inability to follow directions, or have any abdominal wall condition that disallows topical coverage as deemed by the treating physician (e.g. abdominal wound, advanced cellulitis, etc.). We will obtain consent from the patient for incorporating the AGIS device during the inpatient stay. The technical staff will be oriented to the device. However, a physician member of our staff will be available at all times to help position the device if needed. A research coordinator will collect clinical data and enter the data into a secure spreadsheet. Study team members willcollect the following data from patient medical records once patients have consented for the study: Age, Sex, Race/Ethnicity, Body Mass Index (BMI), Abdominal symptoms per chart review, abdominal examination findings per chart review, days in the ICU, days in step down monitoring unit, days in ward, daily vital signs in proximity to the time device is worn, including temperature recordings, respiratory rate recordings, heart rate recordings, blood pressure recordings, and medication usage. Patient data pertaining to their return to bowel function will be abstracted, including: date/time bowel sounds first recorded in chart, date/time first flatus recorded in chart, date/time first bowel movement recorded in chart, date/time of any vomiting episodes, date/time oral diet initiated, amount of diet tolerating, need for placement of nasogastric decompression tubes. Patients will be asked to fill out diaries of their symptoms when possible.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Admission to the SICU

Exclusion Criteria:

* Unable to place sensors on patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical intensive care patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Count of motility events per minute | 1 minute

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars-Sinai Medical Center, Beverly Hills, California, United States

IPD SHARING:
Plan to Share IPD: No